CLINICAL TRIAL: NCT06090279
Title: Feasibility of the Gamification of Incentive Spirometry in Trauma Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: significant delays in acquiring the equipment that was supposed to be loaned for the study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00097144
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-04

CONDITIONS: Thoracic Trauma
Keywords: pulmonary therapies; incentive spirometry; pulmonary complications; pulmonary function; gamification

STUDY DESIGN:
Intervention Model Description: a minimum of 3 rounds of game usage in the Trauma Intensive Care Unit (TICU). Each patient will receive at least 2 sessions per day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OmniFlow Breathing Therapy BioFeeback System (Experimental): This system is a FDA approved healthcare gaming system that is used for patients who have difficulty breathing and allows the patients to participate in breathing exercises for pulmonary rehab.
  Interventions: Device: OmniFlow Breathing Therapy BioFeeback System

INTERVENTIONS:
Device: OmniFlow Breathing Therapy BioFeeback System — FDA approved healthcare gaming system that is used for patients who have difficulty breathing and allows the patients to participate in breathing exercises for pulmonary rehab. Each game usage itself is expected to last 15-20 minutes.
  Other Names: healthcare gaming

SUMMARY:
Gamification may be one solution that can increase the compliance in the use of devices like incentive spirometry.

DETAILED DESCRIPTION:
Recently, there has been much interest in the gamification of healthcare, such as virtual incentive spirometry gaming. Several studies have examined the addition of gamification e.g. virtual incentive spirometry devices. There is a paucity of data regarding the gamification of incentive spirometry, and there is no data involving trauma patients. Previous studies have enrolled either healthy volunteers or patients with specific lung pathology. This study to assess the safety, feasibility and efficacy of respiratory interventions in chest trauma patients using a therapeutic gamification platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if informed consent can be obtained from patient themselves and first session of incentive spirometry gamification can be performed within 48 hours of Trauma Intensive Care Unit (TICU) admission
* Adult patients (≥ 18 years of age) in the TICU with rib fractures or flail segment or a sternal fracture

Exclusion Criteria:

* Trauma patients in the TICU who are mechanically ventilated or requiring bilevel positive airway pressure (BiPAP)
* Glasgow Coma Scale (GCS) < 15, at the time of enrollment
* Facial fractures precluding the use of incentive spirometry
* Any organ injury that precludes use of respiratory therapies in the clinical judgement of the clinical team
* Patients who are expected to be transferred out of the TICU or discharged from the TICU in the next 24 hours based on treating physicians judgment
* Patients who are transitioning to palliative care or expected to die in the next 48 hours based on treating physician's judgment will not be included
* Patients unable to consent for themselves
* Patients unable to use the mouthpiece of the Omniflow system, and those who have visual or hearing impairments that could limit their ability to evaluate the games

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number screened and eligible compared to patient that consented to project | up to 6 months
  Number screened and eligible compared to patient that consented to project
Number of sessions attempted, completed and aborted including the time spent in successful intervention | up to 6 months
  Number of sessions attempted, completed and aborted including the time spent in successful intervention
Reasons for aborting a session related to patient factors, staffing factors, technology factors | up to 6 months
  Enter the results according to the reason
  The Session will be terminated if one or more of the following occurs:
  * Sustained Pain Score >8/10
  * Increase in oxygen requirements by more than 2L/min or hypoxia to less than 92% during the intervention or need for escalation of an oxygen supplementation device
  * Sustained Heart Rate >110 beats per minute, new cardiac arrhythmia or respiratory rate >30 per minute
  * Cyanosis, pallor, or new onset confusion
  * Refusal to continue by choice, reduced engagement in game, adverse symptoms related to dyspnea, pain or discomfort related to the intervention
  * These safety measures are vital sign derangements or signs/symptoms that predict threat to the patient's health
  * Sessions unable to be performed after enrollment due to lack of personnel
  * Failure of intervention device to work, failure of accompanying gamification platform to work
Number of days spent in Intensive Care Unit (ICU) | up to 6 months
  Number of days spent in Intensive Care Unit (ICU)
Number of Subjects readmitted to the ICU for pulmonary complications | up to 6 months
  Number of Subjects readmitted to the ICU for pulmonary complications

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Sarwal, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No